CLINICAL TRIAL: NCT04350827
Title: Platelet-rich Plasma Versus Platelet-rich Plasma Plus Concentrated Insulin-like Growth Factor for Patellar Tendinosis: a Randomized Comparative Trial
Brief Title: PRP vs PRP Plus IGF for Patellar Tendinosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Michael Baria, Assistant Professor, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2019H0437
Record Dates: First submitted 2020-04-15; First posted 2020-04-17 (Actual); Results first posted 2023-10-30 (Actual); Last update posted 2023-10-30 (Actual); Status verified 2023-10

CONDITIONS: Tendinopathy; Patellar Ligament; Platelet-Rich Plasma
MeSH Terms: conditions — Tendinopathy

STUDY DESIGN:
Intervention Model Description: Double blinded randomized comparative trial.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Platelet Rich Plasma (Active Comparator): Procedure will be carried out with excellent sterile technique. 54ml of whole blood will be drawn. 54ml will be processed by centrifugation using the GPS III system (Zimmer Biomet, Warsaw, IN) and 1 ml will undergo a complete blood count (for a baseline comparison to determine the fold increase in platelets). The resultant PRP (5ml) will be injected (after 5ml 1% lidocaine has been injected into the skin for comfort) into the patellar tendon using ultrasound guidance to accurately direct the injection to the site of the tendon abnormality. The patient will rest after the injection for 15 minutes and then be dismissed.
  Interventions: Device: Platelet Rich Plasma
- Platelet Rich Plasma plus IGF (Active Comparator): The PRP preparation and blood draw will be identical to the above. 55ml of whole blood will be drawn (1ml will undergo a CBC and the remaining 54ml will be used to make PRP). In addition to preparing the PRP, the resultant PPP (instead of discarding it) will be placed into the Plasmax device (Zimmer Biomet, Warsaw, IN) and concentrated via a second centrifugation cycle. The plasmax concentrate (concentrated IGF) will be added to the PRP (3ml of PRP + 2ml of plasmax concentrate for a total of 5ml) and then will be injected (after 5ml 1% lidocaine has been injected into the skin for comfort) under ultrasound guidance followed by the same rest period.
  Interventions: Device: Platelet Rich Plasma plus IGF

INTERVENTIONS:
Device: Platelet Rich Plasma — Platelet rich plasma injection into patellar tendon
  Arms: Platelet Rich Plasma
Device: Platelet Rich Plasma plus IGF — Platelet rich plasma plus IGF injection into patellar tendon
  Arms: Platelet Rich Plasma plus IGF

SUMMARY:
The purpose of this study is to compare two different platelet-rich plasma (PRP) injections for patellar tendinosis.

Aim: To perform a randomized, double blinded study comparing the clinical effect of PRP versus PRP + concentrated insulin-like growth factor (IGF) in patients with patellar tendinosis.

DETAILED DESCRIPTION:
Introduction/Background:

Patellar tendinosis is a frustrating ailment commonly encountered in sports medicine. Treating this condition continues to be a significant challenge for sports medicine physicians. The tendinosis lesion is characterized by collagen disorganization and increased ground substance. One method of treating this problem is using platelet rich plasma (PRP), which is a concentration of platelets from the patient's own blood that provides a high dose of growth factors aimed at stimulating tendon healing. These injections have been used extensively to treat many tendon disorders including patellar tendinosis. Several studies have demonstrated the safety and efficacy of using PRP to treat patellar tendinosis.

One growth factor that is known to be helpful in tendon healing is insulin-like growth factor (IGF). However, IGF is not found in PRP but rather in the free plasma that is spun off during the PRP processing. This free plasma or platelet poor plasma (PPP) is typically discarded but it is a known source of IGF. We have shown that concentrating PPP in the FDA cleared Plasmax device yields an increased concentration of insulin-like growth factor (IGF). Local IGF injections into the patellar tendon have demonstrated improved tendon healing, but the effect on clinical outcomes has never been studied in a controlled fashion.

Research Design: Double blinded randomized comparative trial.

Detailed Study Procedures: 38 patients will be randomly assigned to a treatment arm. 19 patients will receive platelet rich plasma (PRP) and 19 patients will receive PRP plus concentrated IGF. Patient will be blinded to their treatment, but treatment team will not. PRP will be prepared according to standard sterile procedures out of view of the patient to ensure patients are adequately blinded. The injecting physician will not be blinded to randomization scheme.

ELIGIBILITY:
Inclusion Criteria:

* >6 weeks of symptomatic patellar tendinosis
* unilateral or bilateral
* 18 yrs of age or older
* active in sport and exercise at least 3x / week
* able to take time away from sport (for healing and rehabilitation phase after procedure)
* failed at least 6 weeks of guided rehabilitation (under the supervision of either a certified athletic trainer or physical therapist)
* minimum Tegner activity level of 4

Exclusion Criteria:

* Steroid injection in target knee in the last 3 months
* PRP in the target knee in the last 6 months
* No other cellular treatments in index knee (bone marrow, amniotic suspensions) last 1 year
* Participation in any experimental device or drug study within 1 year before screening visit
* Oral or IM steroids for last 3 months
* Dry needling of patellar tendon in last 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2020-02-25 (Actual); Primary Completion 2021-10-16 (Actual); Study Completion 2021-10-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Baria, MD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University Sports Medicine Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Andriolo L, Altamura SA, Reale D, Candrian C, Zaffagnini S, Filardo G. Nonsurgical Treatments of Patellar Tendinopathy: Multiple Injections of Platelet-Rich Plasma Are a Suitable Option: A Systematic Review and Meta-analysis. Am J Sports Med. 2019 Mar;47(4):1001-1018. doi: 10.1177/0363546518759674. Epub 2018 Mar 30. PMID 29601207
- [Background] Charousset C, Zaoui A, Bellaiche L, Bouyer B. Are multiple platelet-rich plasma injections useful for treatment of chronic patellar tendinopathy in athletes? a prospective study. Am J Sports Med. 2014 Apr;42(4):906-11. doi: 10.1177/0363546513519964. Epub 2014 Feb 11. PMID 24519184
- [Background] Cole BJ, Karas V, Hussey K, Pilz K, Fortier LA. Hyaluronic Acid Versus Platelet-Rich Plasma: A Prospective, Double-Blind Randomized Controlled Trial Comparing Clinical Outcomes and Effects on Intra-articular Biology for the Treatment of Knee Osteoarthritis. Am J Sports Med. 2017 Feb;45(2):339-346. doi: 10.1177/0363546516665809. Epub 2016 Oct 21. PMID 28146403
- [Background] Dragoo JL, Wasterlain AS, Braun HJ, Nead KT. Platelet-rich plasma as a treatment for patellar tendinopathy: a double-blind, randomized controlled trial. Am J Sports Med. 2014 Mar;42(3):610-8. doi: 10.1177/0363546513518416. Epub 2014 Jan 30. PMID 24481828
- [Background] Dupley L, Charalambous CP. Platelet-Rich Plasma Injections as a Treatment for Refractory Patellar Tendinosis: A Meta-Analysis of Randomised Trials. Knee Surg Relat Res. 2017 Sep 1;29(3):165-171. doi: 10.5792/ksrr.16.055. PMID 28854761
- [Background] Filardo G, Kon E, Della Villa S, Vincentelli F, Fornasari PM, Marcacci M. Use of platelet-rich plasma for the treatment of refractory jumper's knee. Int Orthop. 2010 Aug;34(6):909-15. doi: 10.1007/s00264-009-0845-7. Epub 2009 Jul 31. PMID 19641918
- [Background] Hansen M, Boesen A, Holm L, Flyvbjerg A, Langberg H, Kjaer M. Local administration of insulin-like growth factor-I (IGF-I) stimulates tendon collagen synthesis in humans. Scand J Med Sci Sports. 2013 Oct;23(5):614-9. doi: 10.1111/j.1600-0838.2011.01431.x. Epub 2012 Jan 31. PMID 22288768
- [Background] Ionita CR, Troillet AR, Vahlenkamp TW, Winter K, Brehm W, Ionita JC. Comparison of humoral insulin-like growth factor-1, platelet-derived growth factor-BB, transforming growth factor-beta1, and interleukin-1 receptor antagonist concentrations among equine autologous blood-derived preparations. Am J Vet Res. 2016 Aug;77(8):898-905. doi: 10.2460/ajvr.77.8.898. PMID 27463555
- [Background] Molloy T, Wang Y, Murrell G. The roles of growth factors in tendon and ligament healing. Sports Med. 2003;33(5):381-94. doi: 10.2165/00007256-200333050-00004. PMID 12696985
- [Background] Muir SM, Reisbig N, Baria M, Kaeding C, Bertone AL. The Concentration of Plasma Provides Additional Bioactive Proteins in Platelet and Autologous Protein Solutions. Am J Sports Med. 2019 Jul;47(8):1955-1963. doi: 10.1177/0363546519849671. Epub 2019 May 24. PMID 31125271
- [Background] Patel S, Dhillon MS, Aggarwal S, Marwaha N, Jain A. Treatment with platelet-rich plasma is more effective than placebo for knee osteoarthritis: a prospective, double-blind, randomized trial. Am J Sports Med. 2013 Feb;41(2):356-64. doi: 10.1177/0363546512471299. Epub 2013 Jan 8. PMID 23299850
- [Background] Scott A, LaPrade RF, Harmon KG, Filardo G, Kon E, Della Villa S, Bahr R, Moksnes H, Torgalsen T, Lee J, Dragoo JL, Engebretsen L. Platelet-Rich Plasma for Patellar Tendinopathy: A Randomized Controlled Trial of Leukocyte-Rich PRP or Leukocyte-Poor PRP Versus Saline. Am J Sports Med. 2019 Jun;47(7):1654-1661. doi: 10.1177/0363546519837954. Epub 2019 Apr 30. PMID 31038979
- [Background] Smith PA. Intra-articular Autologous Conditioned Plasma Injections Provide Safe and Efficacious Treatment for Knee Osteoarthritis: An FDA-Sanctioned, Randomized, Double-blind, Placebo-controlled Clinical Trial. Am J Sports Med. 2016 Apr;44(4):884-91. doi: 10.1177/0363546515624678. Epub 2016 Feb 1. PMID 26831629
- [Background] Vetrano M, Castorina A, Vulpiani MC, Baldini R, Pavan A, Ferretti A. Platelet-rich plasma versus focused shock waves in the treatment of jumper's knee in athletes. Am J Sports Med. 2013 Apr;41(4):795-803. doi: 10.1177/0363546513475345. Epub 2013 Feb 13. PMID 23408591

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 14 participants were consented to participate. All met inclusion/exclusion criteria and were randomized.
Period: Overall Study
Arm/Group | Platelet Rich Plasma | Platelet Rich Plasma Plus IGF
Started | 6 | 8
6 Months | 5 | 6
Completed | 5 | 6
Not Completed | 1 | 2
Not completed — Lost to Follow-up | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Platelet Rich Plasma | Platelet Rich Plasma Plus IGF | Total
Number analyzed (Participants) | 6 | 8 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 35 (14) | 35 (10) | 35 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 4
  Male | 5 | 5 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 6 | 7 | 13
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
VISA-P [Mean (Standard Deviation); unit: units on a scale] — Victorian institute of sport assessment scale for patellar tendinopathy [VISA-P] is a self-administered questionnaire consisting of 8 items; 6 are used to evaluate pain levels or disability in daily activities and special functional tests and 2 provide information regarding ability to play sport. The maximum score possible is 100 points and represents an asymptomatic athlete who can fully engage iin sports. The theoretical minimum score is 0 points.
  units on a scale | 43.6 (18.5) | 45.9 (12.5) | 44.9 (14.8)

OUTCOME MEASURES:

1. Primary Outcome: Victorian Institute of Sport Assessment-patellar Tendon (VISA-P)
Description: Victorian Institute of sport assessment scale for patellar tendinopathy [VISA-P] is a self-administered questionnaire consisting of 8 items; 6 are used to evaluate pain levels or disability in daily activities and specific functional tests and 2 provide information regarding ability to play sport. The maximum score possible is 100 points and represents an asymptomatic athlete who can fully engage in sports. The theoretical minimum is 0 points.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Platelet Rich Plasma | Platelet Rich Plasma Plus IGF
Number analyzed (Participants) | 5 | 6
units on a scale | 66.4 (17.8) | 78.2 (15.3)
Statistical Analysis 1: Comparison: Platelet Rich Plasma vs Platelet Rich Plasma Plus IGF; Test type: Superiority; p = 0.433, ANOVA

2. Secondary Outcome: Visual Analog Scale-Pain
Description: The Visual Analog Scale (VAS) measures pain intensity. The VAS consists of a 10cm line, with two end points representing 0 ('no pain') and 10 ('pain as bad as it could possibly be').
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Platelet Rich Plasma | Platelet Rich Plasma Plus IGF
Number analyzed (Participants) | 5 | 6
units on a scale | 2.38 (2.82) | 1.30 (2.07)

3. Secondary Outcome: Tegner Activity Scale
Description: The Tegner activity scale is a one-item score that grads activity based on work and sports activities on a scale of 0 to 10. Zero represents disability because of knee problems and 10 athlete participating in competitive sports.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Platelet Rich Plasma | Platelet Rich Plasma Plus IGF
Number analyzed (Participants) | 5 | 6
units on a scale | 5.8 (1.9) | 6.5 (0.8)

4. Secondary Outcome: Blazina Classification
Description: Classification scale for functional limitations associated with patellar tendinitis. Stage 1: Pain after sports activity, Stage 2: Pain at the beginning of sports activity, disappearing with warm-up and sometimes reappearing with fatigue, Stage 3: Pain at rest and during activity; inability to participate in sports, Stage 4: Rupture of the patellar tendon
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Platelet Rich Plasma | Platelet Rich Plasma Plus IGF
Number analyzed (Participants) | 5 | 6
Participants
  Stage 1 | 4 | 5
  Stage 2 | 0 | 1
  Stage 3 | 1 | 0
  Stage 4 | 0 | 0

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Platelet Rich Plasma | Platelet Rich Plasma Plus IGF
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/6
Other Adverse Events (participants affected / at risk) | 0/5 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-06-02): https://cdn.clinicaltrials.gov/large-docs/27/NCT04350827/Prot_SAP_000.pdf
  • Informed Consent Form (2020-01-15): https://cdn.clinicaltrials.gov/large-docs/27/NCT04350827/ICF_001.pdf